CLINICAL TRIAL: NCT07221435
Title: Microlearning-Based Health Education to Enhance Ambulatory Surgery Patients' Knowledge Retention, Self-efficacy, and Quality of Postoperative Recovery
Brief Title: Microlearning-Based Health Education for Ambulatory Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Adonis Hijaz, MD, Vice Chairman, Department of Urology, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20251195
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Microlearning
Keywords: patient education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microlearning Group (Experimental): Participants in this group will complete the pre-education survey, then they will receive the microlearning education, and complete the post-education survey.
  Interventions: Behavioral: Microlearning education

INTERVENTIONS:
Behavioral: Microlearning education — Participants will receive the link to a technology-based education module. There will be 10 modules and the participant can complete the modules at their own pace.

SUMMARY:
This study is being conducted to explore how microlearning-based health education can improve patients' knowledge, self-confidence in managing their care (self-efficacy), and overall recovery after same-day surgery. Ambulatory surgeries, such as vaginal hysterectomies and mid-urethral sling procedures, are becoming more common because they typically lead to better outcomes and shorter recovery times than inpatient surgeries. Microlearning has been effective in improving knowledge and confidence in other healthcare settings, but is not yet well studied for surgical patients. A total of 50 participants will be enrolled in the study at the University Hospitals. Participants will be patients scheduled for either a mid-urethral sling procedure or a vaginal hysterectomy, and they will complete pre- and post-education surveys as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for the ambulatory mid-urethral sling procedures for stress urinary incontinence OR ambulatory vaginal hysterectomy for uterine prolapse
* Aged 18 to 80
* Able to access technology (mobile phone, computer, tablet, or iPad)
* Demonstrate sufficient proficiency in English to read, write, speak, and understand instructions without the need for translation or interpretation.

Exclusion Criteria:

* Prior experience with ambulatory surgery in the past year
* Diagnosed with Cognitive disorders of dementia or Alzheimer's
* Blindness
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge score as measured by the knowledge test. | Baseline, Post Education (within 2 weeks after surgery)
  The knowledge test was developed in collaboration with both physicians and nursing experts. The test was created to align with the educational objectives and content delivered during the intervention. The test consists of 15 multiple-choice items, with each item carrying a score of 1. The total score is 15, with higher scores indicating a greater level of knowledge. A higher score on the post-test indicates greater retention of knowledge.
Change in Self-Efficacy as measured by the Self-care Self-Efficacy Scale (SCSES) | Baseline, Post Education (within 2 weeks after the surgery)
  The Self-Care Self-Efficacy Scale (SCSES): The instrument consists of 10 items designed to assess self-efficacy related to self-care. Responses are rated on a scale from 1 to 5. The total scores range from 0 to 100, with higher scores indicating greater self-efficacy.
Quality of Postoperative Recovery as measured by the Post-discharge Surgical Recovery (PSR). | Post Education ( within 2 weeks after surgery)
  The PSR is a self-report tool to assess patients' perceived recovery. The PSR consists of 13 items that measure various aspects of recovery. Each item is presented on a visual analogue scale from 0 to 10, with patients circling a number that reflects their response. Scores for each aspect range from 0 to 100, with higher scores indicating better recovery.

SECONDARY OUTCOMES:
The acceptability of the intervention as measured by the Acceptability of Intervention Measure (AIM) | Post Education (within 2 weeks after surgery)
  The AIM consists of 4 items with 5-point ordinal response options from "completely disagree" (1), "Disagree" (2), "Neither Agree nor Disagree" (3), "Agree" (4), and "Completely Agree" (5). The total score is the sum of all items and ranges from 1 to 20. The higher score indicates greater acceptability.
The feasibility of the intervention as measured by the Feasibility of Intervention Measure (FIM). | Post Education (within 2 weeks after surgery)
  The FIM consists of 4 items with 5-point ordinal response options from "completely disagree" (1), "Disagree" (2), "Neither Agree nor Disagree" (3), "Agree" (4), and "Completely Agree" (5). The total score is the sum of all items and ranges from 1 to 20. The higher score indicates greater feasibility.
The appropriateness of the intervention as measured by the Intervention Appropriateness Measure (IAM) | Post Education (within 2 weeks after surgery)
  The IAM consists of 4 items with 5-point ordinal response options from "completely disagree" (1), "Disagree" (2), "Neither Agree nor Disagree" (3), "Agree" (4), and "Completely Agree" (5). The total score is the sum of all items and ranges from 1 to 20. The higher score indicates greater appropriateness.
Number of times the modules were visited as measured by the usage log | Post education ( 2 weeks after surgery)
  The usage log is displayed in the statistics dashboard of the microlearning education modules. This will include metrics of the number of times the educational modules are opened.
Number of modules completed as measured by the modules log. | Post education ( 2 weeks after surgery)
  The number of module completions is displayed in the statistics dashboard of the microlearning education modules. This will include metrics of the number of module completions.
The satisfaction level of the intervention implementation as measured by a 4-point Likert scale. | Post Education (within 2 weeks after surgery)
  The questionnaire includes: "How satisfied are you with the overall Microlearning-based health education?" The Likert scale ranges from 1 to 4. A total score ranges from 1 to 4. A higher score indicates a higher level of satisfaction.
The recommendation likelihood of the intervention as measured by a 4 point Likert scale | Post Education (within 2 weeks after surgery)
  The questionnaire includes:"How likely will you recommend this Microlearning-based health education to others? The Likert scale ranges from 1 to 4. A total score ranges from 1 to 4. A higher score indicates a greater recommendation likelihood of the intervention.
Number of services used after discharge as measured by patient self-report. | Post Education ( within 2 weeks after surgery)
  The number of services used after discharge is measured by the total number of patient-reported clarification calls, emergency room visits, and hospital admissions after discharge.
Cognitive Status as measured by the Mini-Cog© | Baseline
  The Mini-Cog is a brief cognitive screening tool used to assess cognitive impairment. The instrument consists of two components: a three-item recall task and a clock-drawing task. The recall task scores range from 0 to 3. The scoring for clock drawing consists of either 2 or 0 points. The cumulative possible total score ranges from 0 to 5. A total score falling within the range of 0 to 2 points suggests a heightened probability of cognitive impairment warranting further investigation, while a score between 3 to 5 points indicates a low likelihood of cognitive impairment
Health Literacy as measured by the Short Assessment of Health Literacy (SAHL) | Baseline
  The Short Assessment of Health Literacy-Spanish and English (SAHL) is a measure of individuals' health literacy. In administering this assessment, individuals are presented with 18 test terms, one at a time. Scoring for the SAHL includes one point for each correct answer, determined by both correct pronunciation and accurate association with the test item. The total score is 18, with a score between 0 and 14 suggesting low health literacy.
eHealth Literacy as measured by the eHealth Literacy Scale (eHEALS) | Baseline
  eHEALS consists of an 8-item scale measured on a 5-point Likert scale, ranging from 1 to 5. The items assessed an individual's knowledge of online health information resources and their confidence in finding, evaluating, and using this information to make informed health decisions. The eHEALS scores, ranging from 8 to 40, indicate perceived eHealth literacy, with higher scores reflecting greater eHealth literacy and lower scores indicating lesser eHealth literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Adonis Hijaz, MD, Principal Investigator — University Hospitals; Sutthinee Thorngthip, MSN, Principal Investigator — Case Western Reserve University, Frances Payne Bolton School of Nursing
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No